CLINICAL TRIAL: NCT00284336
Title: An Open Label Phase II Trial to Investigate the Cardiac Effects of Pegylated Liposomal Doxorubicine (Caelyx) in Elderly Breast Cancer Patients With New Imaging and Biochemical Techniques.
Brief Title: Caelyx Adjuvant in Elderly Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, prof. dr. Hans Wildiers, adjunct head of clinic, Universitaire Ziekenhuizen KU Leuven
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-002995-13; S28720 UZ KUL
Record Dates: First submitted 2005-12-23; First posted 2006-01-31 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Breast Cancer; Elderly
Keywords: breast cancer; elderly; adjuvant chemotherapy; Caelyx
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin; Cyclophosphamide

INTERVENTIONS:
Drug: Caelyx
  Other Names: liposomal doxorubicin
Drug: endoxan
  Other Names: cyclophosphamide

SUMMARY:
This is an open label Phase II study in elderly patients (65y or older) with early breast cancer who are candidate for adjuvant chemotherapy. A scheme with liposomal doxorubicin (Caelyx) and cyclophosphamide (endoxan) will be used. The aim is to study the cardiac effects of liposomal doxorubicin with new non-invasive techniques, ie strain rate imaging, classical echocardiography, and special blood tests measuring troponin I and BNP.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven early breast cancer requiring adjuvant chemotherapy according to the treating physician (lymph node positive or other features of high risk according to St-Gallen criteria).
* Age > 65 years
* Normal cardiac function (assessment of LVEF by MUGA scan or echocardiography above the lower limit of normal for the institution).
* Performance status 0 to 2 (WHO scale)
* The determination of ER and PgR is mandatory (immunohistochemical methods required; ER and/or PgR positivity is defined as > 1% of positive cells). Also determination of Her2neu is mandatory, either by immunohistochemistry or by FISH
* Adequate organ function (as defined by neutrophils > 1.5 x109/L, Platelets > 100 x 109/L, Hemoglobin > 10 g/dl, total bilirubin > 1.5 UNL, ASAT (SGOT) and ALAT (SGPT) > 1.5 UNL, alkaline phosphatase > 2.5 UNL, creatinine > 1.5 mg/dl (150 µmol/L)
* Complete staging work-up within 2 months prior to registration. All patients will have bilateral mammography, chest X-ray (PA and lateral) and/or CT-scan, abdominal ultrasound and/or CT scan, bone scan. In case of positive bone scan suspicious for metastases, bone X-ray (or bone CT-scan on spinal hot spots) is mandatory to rule out the possibility of metastatic disease. Other tests may be performed as clinically indicated.
* Patients must be accessible for treatment and follow-up.
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Before patient registration/randomization, written informed consent must be given according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

* Metastatic disease (M1)
* Prior systemic anticancer therapy for breast cancer (chemotherapy, hormone therapy of immunotherapy)
* Prior radiation therapy for breast cancer.
* Pre-existing motor or sensory neurotoxicity of a severity > grade 2 by NCI criteria.
* Serious illness or medical condition:

  * Congestive heart failure or unstable angina pectoris, previous history of myocardial infarction within 1 year from study entry, uncontrolled hypertension or high-risk uncontrolled arrythmias
  * History of significant neurological or psychiatric disorders that would prohibit the understanding and giving of informed consent.
  * Active uncontrolled infection
  * Active peptic ulcer, unstable diabetes.
* Past (less than 5 years) or current history of other neoplasm except for curatively treated basal cell skin cancer or in situ carcinoma of the cervix.
* Concurrent treatment with hormonal replacement therapy: this treatment should be stopped at least 15 days before study entry
* Concurrent treatment with other experimental drugs. No participation in another clinical trial with any investigational not marketed drug within 30 days prior to study entry.
* Concurrent treatment with any other anti-cancer therapy.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 16
Dates: Start 2006-01; Study Completion 2007-04

PRIMARY OUTCOMES:
Investigate the effect on cardiac strain rate imaging (SRI) of Caelyx
The relation between cardiac SRI and classical ejection fraction measurement.
The relation between strain rate and blood markers such as troponin-I and BNP

SECONDARY OUTCOMES:
To assess the tolerability of Caelyx containing regimens in elderly breast cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: hans wildiers, MD PhD, Principal Investigator — UH gasthuisberg Leuven
Locations (2):
- Belgium (2):
  - UZ gent, Ghent
  - UH gasthuisberg, Leuven